CLINICAL TRIAL: NCT02009176
Title: The Prospective, Randomized Case-control(RCT) Research of Laparoscope Anatomical and Aon-anatomical Hepatectomy Treat HCC
Brief Title: Laparoscope Anatomical and Aon-anatomical Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shuguo Zheng, MD (Other)
Responsible Party: Sponsor-Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG003; Zhengshuguo (Registry Identifier: Zhengshuguo)
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Laparoscopic; Aon-anatomical hepatectomy; Anatomical hepatectomy; Micrometastases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Micrometastasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscop Anatomical Hepatectomy (Experimental): Total laparoscopic anatomical hepatectomy were performed, combined with cholecystectomy when necessary. The intraoperative ultrasound, hepatic segmental staining were used selectively.
  Interventions: Procedure: Laparoscopic Anatomical Hepatectomy
- Laparoscope Aon-anatomical Hepatectomy (Active Comparator): Total laparoscopic aon-anatomical hepatectomy were performed, combined with cholecystectomy when necessary. The intraoperative ultrasound or hepatic segmental staining will be used to ensure the tumour was completely resected.
  Interventions: Procedure: Laparoscopic Aon-anatomical Hepatectomy

INTERVENTIONS:
Procedure: Laparoscopic Anatomical Hepatectomy — We let the 110 patients divide into A, B groups randomly who are meet the inclusion criteria .Group A is Laparoscopic Anatomical Hepatectomy: Anatomy the corresponding liver segment pedicle and hepatectomy along the Glisson fiber sheath
  Arms: Laparoscop Anatomical Hepatectomy
Procedure: Laparoscopic Aon-anatomical Hepatectomy — We let the 110 patients divide into A, B groups randomly who are meet the inclusion criteria .Group B is Laparoscopic Aon-anatomical Hepatectomy:1 to 2 cm along the edge of the tumor complete hepatectomy
  Arms: Laparoscope Aon-anatomical Hepatectomy

SUMMARY:
The purpose of this study is to compare short-term and long-term efficacy of two surgical methods by laparoscopic hepatectomy, and provide the evidence for the choice of surgical method from the pathology and cytology.

DETAILED DESCRIPTION:
Background:Hepatocellular carcinoma is the world's most common and most malignant tumor, accounting for more than 90% of primary liver cancer, the incidence ranked fifth of malignant tumors in the world. surgery and comprehensive treatment is recognized by the medical profession Surgical approach, including the open HCC hepatectomy and laparoscopic hepatectomy, minimally invasive surgery is the main theme of the 21st century, and laparoscopy as the one of the elements in the field of minimally invasive surgery which carried out more and more in liver surgery, but which one of the two methods to choice to hepatectomy lack of sufficient scientific evidence.The RCT research of laparoscopic anatomical and non-anatomical hepatectomy for HCC has not been reported at home and abroad; Intervention:We let the 110 patients divide into A, B groups randomly who are meet the inclusion criteria .Group A is Laparoscopic Anatomical Hepatectomy: Anatomy the corresponding liver segment pedicle and hepatectomy along the Glisson fiber sheath.Group B is Laparoscopic Aon-anatomical Hepatectomy:1 to 2 cm along the edge of the tumor complete hepatectomy

Results:

1. operation time, intraoperative blood loss, rate of blood transfusion, complications and mortality, postoperative liver function, resection margin, number of micrometastases ,long-term curative effect and survival time were collected and analysed.
2. groups t-test ，univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis ，Kaplan-Meier survival analysis，Log-rank survival curves were used.

ELIGIBILITY:
Inclusion Criteria:

* (1) both male and female, aged 18 to 70; (2) Hepatocellular carcinoma(HCC)diagnosis is clear preoperative; (3) preoperative liver function evaluation: Child-Pugh => B; (4) the lesions can be anatomical hepatectomy,( Indocyanine Green retention rate of 15 minutes) ICGR-15< 20%, the remaining liver volume is sufficient; (5) hepatic single lesions and tumor size between 3-10 cm, does not Invasion the main vein, hepatic artery and vein and major inferior vena cava, did not occur extrahepatic metastasis, and laparoscopic can complete resection; (6) surgery, radiofrequency ablation (RFA), TACE treatment, radiotherapy and chemotherapy have not been implemented (7) voluntary participation in the study, and informed consent.

Exclusion Criteria:

* • (1) age <18 years or> 70 years , pregnant or lactating women; (2) HCC diagnosis is not clear; (3) preoperative liver function evaluation: Child-Pugh C grade; (4) ICGR-15> 20%, the remaining liver volume is insufficient (account for standard liver volume <35%); (5) preoperative tumor has ruptured, or has been undergoing surgery, radiofrequency ablation (RFA), transhepatic arterial chemotherapy and embolization(TACE) or radiotherapy and chemotherapy treatment; (6) preoperative examinations showed multiple (>3)liver lesion or tumor diameter <3 or> 10 cm, a clearly major portal vein, hepatic vein, inferior vena vein tumor thrombus; (7) extrahepatic metastasis; (8) cardio-pulmonary function and other diseases can not tolerate surgery; (9) the patient refused to sign the informed consent form; (10) the tumor has spread and / or lymph node metastasis intraoperative found ; (11) intraoperative found not to be the HCC, such as metastatic hepatic carcinoma, hilar cell carcinoma; (12) Histological examinations showed it is cholangio carcinoma, or mixed liver carcinoma; (13) foreign and Hong Kong, Macao, Taiwan or other areas, estimated that difficult to track, follow-up postoperative

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-03; Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 5 years
  follow-up after the surgery every 2 months, to understand relapse, death, statistics 1 year, 3-year and 5-year survival, disease-free survival, recurrence rate.

SECONDARY OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  hepatic failure,hemorrhage,biliary leakage,ascites,intra-abdominal infection,pleural effusion,pulmonary infection,cardiac insufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Bosch FX, Ribes J, Diaz M, Cleries R. Primary liver cancer: worldwide incidence and trends. Gastroenterology. 2004 Nov;127(5 Suppl 1):S5-S16. doi: 10.1053/j.gastro.2004.09.011. PMID 15508102
- [Background] Kaido T. Recent randomized controlled trials in hepatectomy. Hepatogastroenterology. 2007 Sep;54(78):1825-30. PMID 18019727
- [Background] Man K, Fan ST, Ng IO, Lo CM, Liu CL, Wong J. Prospective evaluation of Pringle maneuver in hepatectomy for liver tumors by a randomized study. Ann Surg. 1997 Dec;226(6):704-11; discussion 711-3. doi: 10.1097/00000658-199712000-00007. PMID 9409569
- [Background] Figueras J, Llado L, Ruiz D, Ramos E, Busquets J, Rafecas A, Torras J, Fabregat J. Complete versus selective portal triad clamping for minor liver resections: a prospective randomized trial. Ann Surg. 2005 Apr;241(4):582-90. doi: 10.1097/01.sla.0000157168.26021.b8. PMID 15798459
- [Background] Kobayashi A, Miyagawa S, Miwa S, Nakata T. Prognostic impact of anatomical resection on early and late intrahepatic recurrence in patients with hepatocellular carcinoma. J Hepatobiliary Pancreat Surg. 2008;15(5):515-21. doi: 10.1007/s00534-007-1293-7. Epub 2008 Oct 4. PMID 18836806
- [Background] Hasegawa K, Kokudo N, Imamura H, Matsuyama Y, Aoki T, Minagawa M, Sano K, Sugawara Y, Takayama T, Makuuchi M. Prognostic impact of anatomic resection for hepatocellular carcinoma. Ann Surg. 2005 Aug;242(2):252-9. doi: 10.1097/01.sla.0000171307.37401.db. PMID 16041216
- [Background] Poon RT, Fan ST, Lo CM, Ng IO, Liu CL, Lam CM, Wong J. Improving survival results after resection of hepatocellular carcinoma: a prospective study of 377 patients over 10 years. Ann Surg. 2001 Jul;234(1):63-70. doi: 10.1097/00000658-200107000-00010. PMID 11420484
- [Background] Zhou XD. Recurrence and metastasis of hepatocellular carcinoma: progress and prospects. Hepatobiliary Pancreat Dis Int. 2002 Feb;1(1):35-41. PMID 14607620
- [Background] Hanazaki K, Kajikawa S, Shimozawa N, Matsushita A, Machida T, Shimada K, Yazawa K, Koide N, Adachi W, Amano J. Perioperative blood transfusion and survival following curative hepatic resection for hepatocellular carcinoma. Hepatogastroenterology. 2005 Mar-Apr;52(62):524-9. PMID 15816471
- [Background] Man K, Ng KT, Lo CM, Ho JW, Sun BS, Sun CK, Lee TK, Poon RT, Fan ST. Ischemia-reperfusion of small liver remnant promotes liver tumor growth and metastases--activation of cell invasion and migration pathways. Liver Transpl. 2007 Dec;13(12):1669-77. doi: 10.1002/lt.21193. PMID 18044786
- [Background] Man K, Lo CM, Xiao JW, Ng KT, Sun BS, Ng IO, Cheng Q, Sun CK, Fan ST. The significance of acute phase small-for-size graft injury on tumor growth and invasiveness after liver transplantation. Ann Surg. 2008 Jun;247(6):1049-57. doi: 10.1097/SLA.0b013e31816ffab6XXX. PMID 18520234
- [Derived] Liao K, Yang K, Cao L, Lu Y, Zheng B, Li X, Wang X, Li J, Chen J, Zheng S. Laparoscopic Anatomical Versus Non-anatomical hepatectomy in the Treatment of Hepatocellular Carcinoma: A randomised controlled trial. Int J Surg. 2022 Jun;102:106652. doi: 10.1016/j.ijsu.2022.106652. Epub 2022 May 4. PMID 35525414